CLINICAL TRIAL: NCT07408076
Title: Sodium Bicarbonate as an Alternative to Potassium Citrate for Kidney Stones
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of California, Davis (Other); Brigham and Women's Hospital (Other); Landspitali University Hospital (Other); University of California, San Diego (Other); Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Principal Investigator, Kymora Scotland, MD, PhD, MD, PhD, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB-24-5580; IRB-24-5580 (Registry Identifier: University of California, Los Angeles IRB)
Record Dates: First submitted 2026-01-16; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Kidney Stones, Urolithiasis, Hypocitraturia; Nephrolithiasis
Keywords: kidney stone; stone; calcium oxalate; calcium phosphate; potassium citrate; sodium bicarbonate; nephrolithiasis
MeSH Terms: conditions — Kidney Calculi; Urolithiasis; Nephrolithiasis; Calculi | interventions — Potassium Citrate; Sodium Bicarbonate

STUDY DESIGN:
Intervention Model Description: 1. Patients with confirmed hypocitraturia identified and enrolled in study
  2. Pre-study medical history and laboratory data will be recorded, and 24 hour urine will be obtained
  3. Set diet will be followed x 48hrs while on first treatment (sodium bicarbonate or potassium citrate; order randomized for 50:50 chance) for at least 1 week
  4. 24 Hour urine performed during 2nd day of set diet
  5. 1 week washout
  6. 1 week use of other medication (sodium bicarbonate or potassium citrate)
  7. Set diet will be followed x 48hrs while on potassium citrate
  8. 24 Hour urine performed during 2nd day of set diet
  9. Change in citrate, pH, and ammonia will be recorded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sodium Bicarbonate -> Potassium Citrate (Experimental): Receives 1 week of sodium bicarbonate, then 1 week of potassium citrate after washout.
  Interventions: Drug: Potassium Citrate; Drug: Sodium Bicarbonate
- Potassium Citrate -> Sodium Bicarbonate (Experimental): 1 week of potassium citrate first, then sodium bicarbonate after a washout.
  Interventions: Drug: Potassium Citrate; Drug: Sodium Bicarbonate

INTERVENTIONS:
Drug: Potassium Citrate — 20 mEq Kcit twice a day (40 mEq daily
Drug: Sodium Bicarbonate — 650 mg sodium bicarbonate twice a day (35.2 mEq daily)

SUMMARY:
Kidney stones affect 1 in every 11 people in the US each year. In patients with kidney stones who are prescribed medications for stone management, only 30.2% are adherent to a medication regime and even fewer, only 13.4 % are adherent with citrate medications.

Prescription potassium citrate can be expensive for many patients, leading to non-compliance. Sodium bicarbonate is a potential medication alternative that is cheaper and can potentially alkalinize the urine and/or decrease the risk of future kidney stones. However, efficacy of alternatives to potassium potassium citrate are not well studied.

This study seeks to evaluate sodium bicarbonate and assess its ability to alkalinize urine in a cohort of patients with kidney stones and compare this to prescription potassium citrate.

DETAILED DESCRIPTION:
Kidney stones affect 1 in every 11 people in the United States each year. A recurrence rate of 50% at 10 years highlights the importance of metabolic management, which has shown to be effective at decreasing the recurrence of stone disease. Specialty guidelines have recommended that clinicians offer pharmacologic therapy to recurrent stone formers. However, among kidney stone patients prescribed medication for stone management, only 30.2% are adherent to a medication regimen and even fewer, only 13.4%, are adherent with citrate medications.

Prescription potassium citrate (Kcit) can be cost-prohibitive for many patients, leading to non-compliance. The combination of the effectiveness of medication with the prohibitory cost of the prescriptions has led to the exploration of treatment alternatives which promise to alkalinize the urine and/or decrease the risk of future kidney stones, including sodium bicarbonate. However, the efficacy of these alternatives in comparison to Kcit are not well studied and often include other alkali equivalents.

A short-term study with limited sample size suggests sodium bicarbonate to be a viable alternative to Kcit. Our goal is to evaluate sodium bicarbonate and assess its ability to alkalinize urine in a cohort of stone-forming patients and compare this to prescription Kcit.

ELIGIBILITY:
Inclusion Criteria:

* Adult >18 years of age
* History of nephrolithiasis
* One 24h urine collections within one year of enrollment with hypocitraturia.
* Patients currently utilizing or considering use of Kcit for stone prevention

Exclusion Criteria:

* Individuals with known metabolic disorders
* Individuals with other known causes of nephrolithiasis
* Anyone who, in the opinion of the PI, is unfit or unsuitable to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in 24-Hour Urinary Citrate Excretion from 24-Hour Urine Collection | 14 days
  Change in 24-hour urinary citrate excretion measured from 24-hour urine collections obtained at baseline and after intervention.
  To determine if sodium bicarbonate is not significantly worse than potassium citrate by more than a clinically acceptable margin of -10
  Unit: mg/day

SECONDARY OUTCOMES:
Change in Urine pH Measured from 24-Hour Urine Collection | 14 days
  Change in urine pH measured from 24 hour urine collections obtained at baseline and after intervention
  units: pH
Change in 24 hour Urinary Ammonia Excretion from 24 Hour Urine Collection | 14 days
  Change in 24 hour urinary ammonia excretion from 24 hour urine collections obtained at baseline and after intervention
  Unit: mmol/day

OTHER OUTCOMES:
Incidence of Side Effects | 14 days
  Number of participants experiencing side effects attributed to the intervention
  Unit: number of participants with ≥1 adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Kymora B Scotland, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (6):
- United States (4):
  - University of California, Los Angeles, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - University of California, San Diego, San Diego, California
  - Brigham & Women's, Boston, Massachusetts
- CHUM, Montreal, Canada
- Landspitali- National University Hospital of Iceland, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results reported in this study, along with the Study Protocol and Statistical Analysis Plan, will be made available to qualified researchers upon request. Interested parties should direct their inquiries and research proposals to KScotland@mednet.ucla.edu. To gain access, requestors will be required to provide a methodologically sound proposal and sign a formal Data Use Agreement (DUA) to ensure participant confidentiality. Data will be available beginning 6 months after the publication of the primary results and will remain accessible for a period of 3 years. The study team will review all requests to determine if the proposed use of the data aligns with the original study's ethical approvals and scientific objectives.
Supporting Information: Study Protocol, SAP
Time Frame: Starting 6 months after publication
  Ending 3 years after publication
Access Criteria: Researchers who submit a research proposal with justified rationale for why they need to access the data along with sound methodological approach, pending approval by the corresponding author. De-identified IPD (ie. baseline characteristics, outcomes, and adverse events) reported from this study will be made available along with study protocol and statistical analysis plan.

REFERENCES:
- [Background] Xue W, Cheng J, Zhao J, Wang L, Peng A, Liu X. Comparison potassium sodium hydrogen citrate with sodium bicarbonate in urine alkalization: a prospective crossover-controlled trial. Int Urol Nephrol. 2023 Jan;55(1):61-68. doi: 10.1007/s11255-022-03387-y. Epub 2022 Oct 19. PMID 36261757
- [Background] Pinheiro VB, Baxmann AC, Tiselius HG, Heilberg IP. The effect of sodium bicarbonate upon urinary citrate excretion in calcium stone formers. Urology. 2013 Jul;82(1):33-7. doi: 10.1016/j.urology.2013.03.002. Epub 2013 Apr 18. PMID 23602798
- [Background] Dauw CA, Yi Y, Bierlein MJ, Yan P, Alruwaily AF, Ghani KR, Wolf JS Jr, Hollenbeck BK, Hollingsworth JM. Factors Associated With Preventive Pharmacological Therapy Adherence Among Patients With Kidney Stones. Urology. 2016 Jul;93:45-9. doi: 10.1016/j.urology.2016.03.030. Epub 2016 Mar 31. PMID 27041472
- [Background] Pearle MS, Goldfarb DS, Assimos DG, Curhan G, Denu-Ciocca CJ, Matlaga BR, Monga M, Penniston KL, Preminger GM, Turk TM, White JR; American Urological Assocation. Medical management of kidney stones: AUA guideline. J Urol. 2014 Aug;192(2):316-24. doi: 10.1016/j.juro.2014.05.006. Epub 2014 May 20. PMID 24857648
- [Background] Pearle MS, Roehrborn CG, Pak CY. Meta-analysis of randomized trials for medical prevention of calcium oxalate nephrolithiasis. J Endourol. 1999 Nov;13(9):679-85. doi: 10.1089/end.1999.13.679. PMID 10608521
- [Background] Barcelo P, Wuhl O, Servitge E, Rousaud A, Pak CY. Randomized double-blind study of potassium citrate in idiopathic hypocitraturic calcium nephrolithiasis. J Urol. 1993 Dec;150(6):1761-4. doi: 10.1016/s0022-5347(17)35888-3. PMID 8230497
- [Background] Ettinger B, Pak CY, Citron JT, Thomas C, Adams-Huet B, Vangessel A. Potassium-magnesium citrate is an effective prophylaxis against recurrent calcium oxalate nephrolithiasis. J Urol. 1997 Dec;158(6):2069-73. doi: 10.1016/s0022-5347(01)68155-2. PMID 9366314
- [Background] Uribarri J, Oh MS, Carroll HJ. The first kidney stone. Ann Intern Med. 1989 Dec 15;111(12):1006-9. doi: 10.7326/0003-4819-111-12-1006. PMID 2688503
- [Background] Scales CD Jr, Smith AC, Hanley JM, Saigal CS; Urologic Diseases in America Project. Prevalence of kidney stones in the United States. Eur Urol. 2012 Jul;62(1):160-5. doi: 10.1016/j.eururo.2012.03.052. Epub 2012 Mar 31. PMID 22498635